CLINICAL TRIAL: NCT05472961
Title: Eye Movement Studies of Visual Search
Brief Title: Eye Movements in Visual Search
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No human participants were required as part of the computational modelling for this experiment during the period of this project. No participants were recruited and no data was collected.
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Thomas J. Palmeri, Distinguished Professor of Psychology, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 140970
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: eye tracker; visual perception

STUDY DESIGN:
Intervention Model Description: Participants are asked to view an array of objects on a computer screen equipped with a noninvasive eye tracker. They are asked to search for a target object among one or more distractor objects and may be asked to respond to a feature of the target object with a key press that was selected via a gaze shift.
Masking Description: Manipulation is within-participant. Participants view multiple visual search arrays in an experimental session. They will be masked with regards to the difficulty and timing manipulations until they experience them on a trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Within Subjects Experimental Design (Experimental): All participants are tested in all conditions.
  Interventions: Behavioral: Target and Stimulus

INTERVENTIONS:
Behavioral: Target and Stimulus — The investigators manipulate the difficulty of search for the target object by manipulating the number of distractor objects and/or the similarity between the target and distractors. The investigators manipulate the difficulty of the decision about a feature by manipulating the similarity of the feature to a criterion. The investigators manipulate the timing of when the decision feature appears on the object relative to the onset of the array and/or the onset of the saccade away from fixation in a gaze-contingent manner.

SUMMARY:
Using a noninvasive eye tracker, the investigators will measure how participants move their eyes to objects arrayed on a computer screen. Participants will be asked to find one element among many.

DETAILED DESCRIPTION:
The investigators measure how quickly and how accurately participants can move their eyes from a central fixation point to a target object arrayed with one or more distractor objects. A noninvasive eye tracker will be used to measure their eye movements. Participants may also be asked to make a decision about a feature of the target they have selected with a key press. Difficulty of the search for the target object and difficulty of the decision about a feature of the target object will be manipulated.

ELIGIBILITY:
Inclusion Criteria:

* Sona System users (open to the public)

Exclusion Criteria:

* participants that fail the Ishihara color vision screening test
* participants with acuity worse than 20/20 with or without correction
* children under 18
* adults over 50

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Eye Tracking Data | During 1-2 hour experimental session
  Saccade Events, Fixation Events, Pupil Size
Response Data | During 1-2 hour experimental session
  Response Time, Error Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified behavioral data will be shared with other investigators upon request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be shared after all analyses and modeling of the data are complete and manuscripts resulting from the research are accepted for publication.
Access Criteria: We will share data with investigators who request (after research using the data are complete).